CLINICAL TRIAL: NCT05841927
Title: Clinical Cohort Study of DHA in Neurodevelopmental Disorders
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: DHA_CHFU
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Autism or Autistic Traits
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASD active (Experimental): Dietary Supplement: Docosahexaenoic acid 200mg DHA once, twice a day
  Interventions: Dietary Supplement: Docosahexaenoic acid supplement
- ASD placebo (Placebo Comparator): Dietary Supplement: Placebo dietary intervention Vitamin D 400IU once, once a day
  Interventions: Dietary Supplement: ASD placebo

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid supplement — Docosahexaenoic acid supplement
  Arms: ASD active
Dietary Supplement: ASD placebo — ASD placebo
  Arms: ASD placebo

SUMMARY:
Neurodevelopmental disorders are a group of developmental disorders, including autism spectrum disorders (ASDs), attention deficit hyperactivity disorder (ADHD) and others, that begin at a developmental stage and severely affect the growth and development of the brain. Autism spectrum disorder (ASD) encompasses a group of neurodevelopmental syndromes characterized by deficits in social interaction and communication as well as repetitive behaviors and restricted interests. There is strong evidence for the involvement of inherited genetic factors in ASD (accounting for at least 80% of the variation in disease risk). There is strong evidence for the involvement of inherited genetic factors in ASD (accounting for at least 80% of the variation in disease risk). According to a meta-analysis, monogenic mutations in SHANK3, which encodes the major postsynaptic density (PSD) scaffolding protein at excitatory glutamatergic synapses, are found in approximately 0.69% of ASD cases and up to 2.12% of all moderate to profound intellectual disability cases. De novo mutations, interstitial deletions, and terminal deletions have been identified in ASD.

Recent studies have shown that children with ASD have significantly lower levels of docosahexaenoic acid (DHA) than those without. Studies have shown that higher DHA intake reduces the risk of schizophrenia, bipolar disorder, depression, anxiety disorder, and conduct disorders. After DHA treatment, most children with ASD showed clinical and biochemical improvements, with increased DHA levels as measured by blood analysis and significant improvements in social scale scores in the supplement group. Moreover, increasing DHA levels in children with ADHD through dietary supplements can improve behavior, attention, literacy, cognitive problems, and working memory function. Therefore, for neurodevelopmental disorders, high DHA intake may be an important component of disease prevention.

DETAILED DESCRIPTION:
For neurodevelopmental disorders, high DHA intake may be an important component of disease prevention. DHA is a safe dietary supplement and is safe for children. Clinical diagnosis and treatments of SHANK, ASD and ADHD were carried out for a long time and a solid foundation for clinical cohort research has accumulated. This study aims to observe the effectiveness of DHA supplementation as an adjuvant therapy for ASD by establishing randomized cohort cases.

ELIGIBILITY:
Inclusion Criteria:

1. Children who were admitted to the Department of Child Care and Developmental Behavior of our hospital and diagnosed as ASD by developmental pediatricians according to the diagnostic criteria of DSM-5.
2. Willing to participate in the study, consume the treatment and perform all measurements including developmental or cognitive testing, blood drawing, anthropometry and questionnaires etc.
3. Informed consent signed by parent or caregiver.

Exclusion Criteria:

1. Children with immune deficiency.
2. Children with major organ malformations (congenital heart disease, nervous system tumors, obvious structural abnormalities of the nervous system, digestive tract malformations, etc.)
3. Have a history of DHA allergy or obvious adverse reactions

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Plasma level concentration of DHA (μg/ml) | 1, 3, 6 months
  Detection and analysis of free fatty acid substances were performed using an Agilent 7890B gas chromatograph system coupled with a Agilent 5977B mass spectrometer.

SECONDARY OUTCOMES:
Change in developmental assessment | 1, 3, 6 months
  Griffiths Mental Development Scales (Griffiths) were conducted by licensed and certified clinicians to assess developmental and cognitive level which is applicable to the children with mental age (not physical age) from 0 to 8.
  The developmental quotient in each zone represents the developmental status of the child. The higher the developmental quotient, the better the child's development.
Change in autism severity assessed by DSM-5 | 1, 3, 6 months
  ASD severity was based on the DSM-5 administrated by certified clinicians. The higher the score, the more severe the symptoms
Change in autism severity | 1, 3, 6 months
  ASD severity was based on the ADOS-2 administrated by certified clinicians. The higher the score, the more severe the symptoms
Change in social adaptation ability | 1, 3, 6 months
  The scales of the Vineland II are organized within a three-domain structure: Communication, Daily Living, and Socialization. This structure corresponds to the three broad domains of adaptive functioning by the American Association of Intellectual and Developmental Disabilities: Conceptual, Practical, and Social. In addition, Vineland II offers a Motor Skills Domain and an optional Maladaptive Behavior Index to provide more in-depth information.
  The higher the score, the better the child's development

CONTACTS AND LOCATIONS:
Overall Officials: Xiu Xu, Principal Investigator — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No